CLINICAL TRIAL: NCT01653288
Title: A Randomized Controlled Trial of "Coping Coach," a Web-based Preventive Intervention for Children
Brief Title: A Trial of "Coping Coach," a Web-based Preventive Intervention for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12-009336; 1R21HD069832-01A1 (NIH)
Record Dates: First submitted 2012-07-25; First posted 2012-07-31 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Stress Disorders, Post Traumatic
MeSH Terms: conditions — Combat Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coping Coach (Experimental): Receive access to Coping Coach online intervention at baseline for use (self-guided, with email reminders) over the next 6 weeks.
  Interventions: Behavioral: Coping Coach
- Coping Coach Waitlist Control (Experimental): Treatment as usual from baseline to 12 week follow-up assessment. Then receive access to Coping Coach intervention after 12 week follow-up for use (self-guided, with email reminders) over the next 6 weeks.
  Interventions: Behavioral: Coping Coach

INTERVENTIONS:
Behavioral: Coping Coach — Coping Coach is a self-guided web-based intervention that utilizes an interactive, developmentally appropriate, game-like format, to provide practical information and teach children adaptive coping strategies. Children are primary users of the intervention, with parent supervision. Modules (20-30 minutes each) can be repeated to solidify skills / learning. The feelings module targets recognition of emotions after potentially traumatic experiences. The appraisals module targets the connection of helpful or unhelpful thoughts to feelings and behavior. The avoidance module targets reducing reliance on avoidance as a (maladaptive) coping response. Promoting social support is folded throughout the intervention. Information will be provided to parents about how to access additional resources and when to get additional professional help.

SUMMARY:
This study will evaluate the impact of a psychosocial intervention, Coping Coach, delivered online to children who have experience an acute medical event.

The core study hypotheses are that children receiving the intervention will (1) endorse fewer maladaptive trauma-related appraisals and (2) demonstrate more adaptive coping (more support-seeking, more cognitive restructuring, less avoidant coping) at a 6-week follow-up, and (3) demonstrate lower severity of post traumatic stress (PTS) symptoms and higher health related quality of life (HRQOL) at 12 week follow-up.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the feasibility and provide an initial evaluation of the efficacy of Coping Coach, a new web-based intervention for children experiencing acute medical events.

The study aims to (1) assess and maximize intervention feasibility, (2) conduct an initial efficacy testing (pilot RCT) for proximal outcomes (appraisals, coping) and subsequent child health outcomes (PTS reactions, HRQOL), and (3) refine the conceptual framework and optimize the intervention effectiveness.

Study Design:

This study will progress in multiple stages:

Pilot study: 20 children experiencing a potentially traumatic medical event will be given the Coping Coach intervention with follow-up at 6 weeks. This pilot will examine initial feasibility, usability, acceptability, and child engagement/ comprehension of the intervention.

Additional Pilot Study (2015): 20 children treated in the ED or admitted to the hospital with injury due to non-family violence will be provided with the Coping Coach intervention. Other inclusion and exclusion criteria, as well as baseline, 6- and 12-week assessments parallel those from the RCT stage described below. This pilot will examine feasibility, engagement, and estimate pre-post changes in key measures in children with violence exposure.

RCT: A wait-list design will compare intervention use with a waitlist control on proximal and child health outcomes at 6, 12, and 18 weeks after baseline enrollment. The Coping Coach intervention will be provided to the waitlist control after the 12 week assessment. 70 children will be enrolled, 35 in each arm. (Assessment of feasibility and engagement will continue in this stage.)

The rest of this CLINICALTRIALS.GOV record describes the RCT (N=72).

The Pilot and RCT combined will help us prepare for rigorous large-scale RCT of Coping Coach.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 8 to 12 years of age
* Child has experienced a potentially traumatic medical event* within the past 2 weeks
* Child's GCS > 12
* Child speaks English well enough to complete the measures and participate in an interview
* Child has access to the Internet and telephone
* Parental/legal guardian informed consent and child assent

Exclusion Criteria:

* Child's current medical condition or cognitive limitations preclude participating in an interview
* Child's acute medical event is due to family violence or suspected child abuse
* Child or parent has been arrested or is subject to legal proceedings related to the index incident
* In the index event, child or parent was a perpetrator of violence (or participant in mutual violence)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Kassam-Adams, PhD, Principal Investigator — Center for Injury Research & Prevention, Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kassam-Adams N, Marsac ML, Kohser KL, Kenardy J, March S, Winston FK. Pilot Randomized Controlled Trial of a Novel Web-Based Intervention to Prevent Posttraumatic Stress in Children Following Medical Events. J Pediatr Psychol. 2016 Jan-Feb;41(1):138-48. doi: 10.1093/jpepsy/jsv057. Epub 2015 Jun 18. PMID 26089554

RESULTS

PARTICIPANT FLOW:
Groups:
- Coping Coach Waitlist Control: Treatment as usual till 12 wk assessment, then access to Coping Coach intervention for use (self-guided, email reminders) over next 6 wks.
  Coping Coach: Coping Coach is a self-guided web-based intervention that utilizes an interactive, developmentally appropriate, game-like format, to provide practical information and teach children adaptive coping strategies. Children are primary users of the intervention, with parent supervision. Modules (20-30 minutes each) can be repeated to solidify skills / learning. The feelings module targets recognition of emotions after potentially traumatic experiences. The appraisals module targets the connection of helpful or unhelpful thoughts to feelings and behavior. The avoidance module targets reducing reliance on avoidance as a (maladaptive) coping response. Promoting social support is folded throughout the intervention. Information will be provided to parents about how to access additional resources and when to get additional professional help.
Period: Overall Study
Arm/Group | Coping Coach | Coping Coach Waitlist Control
Started | 36 | 36
Completed | 26 | 35
Not Completed | 10 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coping Coach | Coping Coach Waitlist Control | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 36 | 72
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (1.5) | 9.8 (1.3) | 9.8 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 21 | 18 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Child race / ethnicity: Black | 12 | 12 | 24
  Child race / ethnicity: White | 21 | 24 | 45
  Child race / ethnicity: Other race / ethnicity | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 36 | 72
Parent education [Count of Participants; unit: Participants]
  Attended or completed high school | 7 | 7 | 14
  Attended college | 20 | 8 | 28
  Completed college or graduate degree | 9 | 21 | 30
Annual household income [Count of Participants; unit: Participants]
  less than $30K | 10 | 6 | 16
  $30K to less than $50K | 8 | 7 | 15
  $50K to less than $75K | 4 | 4 | 8
  $75K to less than $100K | 5 | 4 | 9
  $100K or more | 8 | 15 | 23
  Not reported | 1 | 0 | 1
Type of acute medical event experienced by child [Count of Participants; unit: Participants]
  Appendicitis | 13 | 18 | 31
  Asthma-related | 4 | 2 | 6
  Abdominal pain | 3 | 3 | 6
  Acute joint pain or arthritis | 1 | 3 | 4
  Other acute medical illness | 9 | 6 | 15
  Injury | 6 | 4 | 10
Child's prior trauma exposure [Count of Participants; unit: Participants]
  Any prior trauma: yes | 27 | 25 | 52
  Any prior trauma: no | 9 | 11 | 20
  Prior interpersonal trauma: yes | 7 | 3 | 10
  Prior interpersonal trauma: no | 29 | 33 | 62
  Prior non-interpersonal trauma: yes | 27 | 24 | 51
  Prior non-interpersonal trauma: no | 9 | 12 | 21
Baseline stats for outcome measures [Mean (Standard Deviation); unit: units on a scale] — Child PTSD Symptom Scale (CPSS) measures child posttraumatic stress symptoms, possible range 0-51, high scores = more severe.
  Pediatric Quality of Life Inventory (PedsQL) measures child health-related quality of life, possible range 0-100, high scores = better quality of life.
  How I Coped Under Pressure Scale (HICUPS) measures child avoidance coping strategies, possible range 12-48, high scores = more use of avoidance coping.
  Child Posttraumatic Cognitions Inventory (CPTCI) measures child post trauma cognitive appraisals, possible range 25-100, high scores = more maladaptive appraisals.
  units on a scale
    mean (SD) CPTCI score - maladaptive appraisals | 45.4 (12.1) | 40.5 (11.6) | 43.0 (12.0)
    mean (SD) HICUPS score - avoidance coping) | 32.4 (7.3) | 29.3 (7.4) | 30.9 (7.5)
    mean (SD) CPSS score - traumatic stress severity | 18.4 (11.8) | 13.3 (7.3) | 15.6 (10.1)
    mean (SD) PedsQL score - health quality of life | 78.0 (17.3) | 82.1 (15.8) | 79.9 (16.6)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Coping Coach Online Intervention
Description: Feasibility was measured using automated monitoring data, the number of participants who logged in at least once and the number of participants who completed the entire online intervention are presented here.
Time Frame: 6 weeks
Population: Analyzing usage among all participants who received access (i.e. information on how to sign in) to the Coping Coach online intervention. 28 of 36 in the waitlist control condition completed a 12 week research assessment and then received sign-in information.
Measure: Count of Participants; unit: Participants
Groups:
- Coping Coach: Usage data reported for baseline to week 6
  Receive access to Coping Coach online intervention at baseline for use (self-guided, with email reminders) over the next 6 weeks.
- Coping Coach Waitlist Control: Usage data reported for weeks 12 to 18 (i.e when this arm had access to the online intervention)
  Treatment as usual till 12 wk assessment, then access to Coping Coach intervention for use (self-guided, email reminders) over next 6 wks.
Arm/Group | Coping Coach | Coping Coach Waitlist Control
Number analyzed (Participants) | 36 | 28
Participants
  Logged in / used intervention at least once: yes | 35 | 19
  Logged in / used intervention at least once: no | 1 | 9
  Completed entire online intervention: yes | 19 | 15
  Completed entire online intervention: no | 17 | 13

2. Primary Outcome: Mean Time Spent Using the Intervention
Description: Feasibility was measured using automated monitoring data. Mean time spent using the online intervention, across all sessions, in minutes is reported here.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Coping Coach | Coping Coach Waitlist Control
Number analyzed (Participants) | 36 | 28
minutes | 52.2 (36.9) | 51.5 (30.7)

3. Secondary Outcome: a Preliminary Assessment of the Efficacy of the Intervention
Description: Child PTSD Symptom Scale (CPSS) measures child posttraumatic stress symptoms, possible range 0-51, high scores = more severe.
  Pediatric Quality of Life Inventory (PedsQL) measures child health-related quality of life, possible range 0-100, high scores = better quality of life.
  How I Coped Under Pressure Scale (HICUPS) measures child avoidance coping strategies, possible range 12-48, high scores = more use of avoidance coping.
  Child Posttraumatic Cognitions Inventory (CPTCI) measures child post trauma cognitive appraisals, possible range 25-100, high scores = more maladaptive appraisals.
Time Frame: 6 weeks
Population: descriptive statistics for all randomized participants who completed these measures at 6 week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coping Coach | Coping Coach Waitlist Control
Number analyzed (Participants) | 24 | 34
units on a scale
  mean (SD) CPTCI score - maladaptive appraisals | 45.9 (10.6) | 43.8 (10.5)
  mean (SD) HICUPS score - avoidance coping | 35.4 (7.9) | 31.7 (5.9)
  mean (SD) CPSS score - traumatic stress severity | 13.0 (12.1) | 12.5 (10.0)
  mean (SD) PedsQL score - health quality of life | 75.1 (19.1) | 81.4 (17.5)

4. Secondary Outcome: a Preliminary Assessment of the Efficacy of the Intervention
Description: as for outcome 3
Time Frame: 12 weeks
Population: descriptive statistics for all randomized participants who completed these measures at 12 week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coping Coach | Coping Coach Waitlist Control
Number analyzed (Participants) | 22 | 28
units on a scale
  mean (SD) - CPTCI score - maladaptive appraisals | 39.3 (9.0) | 41.3 (11.5)
  mean (SD) HICUPS score - avoidance coping | 30.6 (9.8) | 31.7 (5.7)
  mean (SD) CPSS score - traumatic stress severity | 13.9 (14.3) | 14.6 (12.0)
  mean (SD) PedsQL score - health quality of life | 86.8 (18.3) | 85.1 (15.1)

5. Other Pre Specified Outcome: Preliminary Assessment of Efficacy of Later Use of the Intervention
Description: as for outcome 3
Time Frame: 18 weeks
Population: reporting on all participants who completed follow-up measures at 18 week. Note that at 12 weeks, those in the waitlist control group who completed the 12 week research assessment (N=28) were given access to the online intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coping Coach | Coping Coach Waitlist Control
Number analyzed (Participants) | 20 | 31
units on a scale
  mean (SD) CPTCI score - maladaptive appraisals | 40.8 (12.6) | 41.1 (11.8)
  mean (SD) HICUPS score - avoidance coping | 33.0 (7.6) | 31.4 (6.9)
  mean (SD) CPSS score - traumatic stress severity | 15.3 (12.5) | 11.0 (10.4)
  mean (SD) PedsQL score - health quality of life | 78.5 (23.4) | 90.4 (11.2)

ADVERSE EVENTS:
Arm/Group | Coping Coach | Coping Coach Waitlist Control
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No